CLINICAL TRIAL: NCT00845923
Title: Phase II Proof of Concept Trial of Civamide Patch in the Treatment of Post-herpetic Neuralgia and Post-incisional Neuralgia
Brief Title: Evaluation of Civamide Patch in Treatment of Postherpetic Neuralgia and Post-Incisional Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WL-1001-04-03
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic neuralgia of at least 6 months
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — zucapsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Civamide Patch 0.015% (Other): All subjects in study will receive the Civamide Patch 0.015%
  Interventions: Drug: Civamide Patch

INTERVENTIONS:
Drug: Civamide Patch — Patch containing Civamide (zucapsaicin) 0.015%, containing 0.210 mg Civamide per patch, applied once a day for four weeks.
  Other Names: zucapsaicin

SUMMARY:
This proof of concept study is designed to evaluate the safety and efficacy of topically administered Civamide Patch for the treatment of moderate to severe daily pain associated with postherpetic neuralgia localized to the trunk, and with localized post-incisional neuropathic pain syndromes on the trunk.

DETAILED DESCRIPTION:
There will be up to approximately 20 evaluable subjects in this open-label study. The study is composed of a 1-week non-treatment Baseline Period (Day -7 to -1), during which subjects will be required to complete a Daily Diary assessing overall pain and sleep interference. The 1-week Baseline Period will be followed by a 4-week Treatment Period, in which subjects will apply the Civamide Patch (0.015%) daily 12 hours per day, for a period of 4 weeks, complete a Daily Diary assessing overall pain and sleep interference, followed by a 2-week Post-Treatment Observation Period. In the course of the study, subjects will visit the clinic a total of five times for physical examinations, vital signs, review of diaries, and distribution and collection of test patches. Efficacy assessment will be the mean change from Baseline Period in efficacy variables during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject healthy other than history of postherpetic neuralgia of at least 6 months after healing of a herpes zoster skin rash.
* Subject must be taking a stable dose of a medication(s) for PHN pain, and be expected to remain on this stable daily dose throughout the study.
* Single, localized area of skin on trunk with PHN, measuring approximately 10 x 14 cm or less.
* Average Daily Pain Score of 4 or higher on 11-point Likert scale during the 7-Day Baseline Period.
* Males or females between 18 to 80 years of age, inclusive.
* Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control throughout study or females of non-childbearing potential. Negative urine pregnancy test must be confirmed at Screening.
* Subject agrees not to begin any new concomitant medications during study.

Exclusion Criteria:

* Subject has area of skin on trunk affected by PHN, greater than an area amendable to treatment by the patch, or exhibits active skin disease, infection, severe erythema, or other compromise in integrity of skin which, could influence or interfere with the evaluation of safety or efficacy.
* Subject has history of frequent headache or other painful conditions (other than that associated with PHN), expected to require more than twice a week additional administration of OTC acetaminophen (≤ 1000 mg total daily dose for pain management).
* Clinical, historical or previous laboratory evidence of significant cardiovascular, renal, gastrointestinal, pulmonary, hepatic, endocrine, neurological, psychological, or other systemic disease that might confound the results of study or pose an additional risk to subject.
* Subject is immunocompromised.
* Use of any restricted medication within given time period prior to Baseline Period and throughout study (See Table 1).
* Females who are pregnant, breast-feeding, or planning to become pregnant during study.
* Subject has a history of alcohol and/or drug abuse within past year.
* Subject has previously participated in a Civamide study.
* Subject has participated in another investigational study, or taken another investigational drug within past 4 weeks.
* Subject received neurolytic or neurosurgical therapy for this or previous episodes of postherpetic neuralgia.
* Known hypersensitivity to or contraindication to use of Civamide (zucapsaicin), capsaicin (Zostrix®, Zostrix-HP®, Axsain®, or related products) or to excipients of clinical formulation.
* If, for any other reason the subject is not deemed to be suitable by Investigator, they should not be enrolled.
* Initiation of a medication, discontinuation of a medication or change in regimen of existing medication(s) or therapies less than required period of stable dosing prior to entering Baseline Period.
* Topical use of any moisturizer or similar products on or near treatment area within 48 hours of Day 1 until after completion of Study on Day 43.
* Topical use of any capsaicin-containing product for 60 days prior to Day 1 until after completion of Study on Day 43.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily Pain Score from the Baseline Period to the Average Daily Pain Score of the last week of the Treatment Period. | Day 29 and Day 43

SECONDARY OUTCOMES:
Average Daily Sleep Score | Change from baseline to other weeks in study

CONTACTS AND LOCATIONS:
Overall Officials: Scott Phillips, M.D., Study Chair — Winston Laboratories
Locations (4):
- United States (3):
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Pain and Rehabilitationi Clinic of Chicago, Chicago, Illinois
  - Michigan Head-Pain and Neurological Institute, Ann Arbor, Michigan
- U.T. Pain Specialist, Etobicoke, Ontario, Canada